CLINICAL TRIAL: NCT03688607
Title: Deploying POKE Within Intermountain Healthcare
Acronym: POKE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IHC IRB #1050915
Record Dates: First submitted 2018-09-25; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Newborn; Infection
Keywords: NICU; POKE; Length of Stay; Infection; Neonates
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- POKE: All babies in NICU at Intermountain Healthcare hospitals
  Interventions: Procedure: There will not be an intervention, rather the investigators will deploy best practices and track POKEs within the healthcare system to evaluate clinical and operational outcomes.

INTERVENTIONS:
Procedure: There will not be an intervention, rather the investigators will deploy best practices and track POKEs within the healthcare system to evaluate clinical and operational outcomes. — There will not be an intervention, rather the investigators will deploy best practices and track POKEs within the healthcare system to evaluate clinical and operational outcomes.

SUMMARY:
To assess the impact of POKE on babies, the investigators will longitudinally track outcomes before and after implementation at Intermountain Healthcare's five NICUs. Process outcomes will include the number of total POKEs per baby and the number of painful POKEs per baby, each measured at both the patient-level and NICU-level. Clinical outcomes will include hospital acquired infections, length of stay, and mortality. Financial outcomes will include total variable costs and backfill rate. The effect of POKE on each of these outcomes will be measured using multivariable regression analysis with appropriate distributional families and interaction terms.

DETAILED DESCRIPTION:
POKE was developed and implemented at Dixie Regional Medical Center's Neonatal Intensive Care Unit (NICU) over the past 10 years to eliminate waste and reduce harm in healthcare. POKE is a combination of a unique culture and process, with a supporting database, that is designed to guide and inform care decisions while minimizing POKEs. The program utilizes an implementation framework, educational materials, electronic health records (EHR), and decision support analytics. POKE's initial deployment showed extremely promising results for Intermountain, which included: (1) eliminating 11,000 POKEs per year (a 50% reduction in overall POKEs), (2) realizing $940,000 per year in cost savings (a 28% reduction of overall cost), (3) reducing length of stay by 2 weeks per average stay (a 21% reduction in length of stay), and (4) eliminating Hospital Acquired Infections (i.e., Central-line Associated Bloodstream Infection and Ventilator-associated Pneumonia), translating into 10 lives saved and a $5.2M savings over a decade. POKE will now be deployed and routinized within all Intermountain Healthcare NICUs and be developed as a commercial product for external customers. To assess the impact of POKE on babies, the investigators will longitudinally track several outcomes before and after implementation at Intermountain NICUs. Process outcomes will include the number of total POKEs per baby and the number of painful POKEs per baby, each measured at both the patient-level and NICU-level. Clinical outcomes will include hospital acquired infections, length of stay, and mortality. Financial outcomes will include total variable costs and backfill rate.

ELIGIBILITY:
Inclusion Criteria:

* All babies in Intermountain Healthcare NICU

Exclusion Criteria:

* None

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Babies admitted to hospital
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of POKEs per baby | 1 October 2018 - 31 May 2019
  The primary outcomes will be the number of total POKEs per baby and the number of painful POKEs per baby. We will assess the impact of POKE on each of these outcomes modeled as counts (ie, generalized Poisson distributions) using multivariable regression adjusting for potential confounders including age, gestational age, interaction terms, and nominal indicators of NICU (to account for baseline heterogeneity across sites).

SECONDARY OUTCOMES:
Infection Rate | 1 October 2018 - 31 May 2019
  Also using multivariable regression, the secondary outcomes will be patient-level indicators, including hospital acquired infection (logistic regression)
Length of Stay | 1 October 2018 - 31 May 2019
  Length of stay (scaled beta regression)
Mortality | 1 October 2018 - 31 May 2019
  Mortality (logistic regression)
Total Variable Cost | 1 October 2018 - 31 May 2019
  Total variable costs (log-linear regression)
Aggregate Backfill Rate | 1 October 2018 - 31 May 2019
  aggregated backfill rate (quasibinomial regression)

CONTACTS AND LOCATIONS:
Overall Officials: R. Erick Ridout, MD, Principal Investigator — Intermountain Health Care, Inc.; Terri Kane, RN, MBA, Study Director — Intermountain Health Care, Inc.; Brad Isaacson, PhD, MBA, MSF, Study Director — Intermountain Health Care, Inc.
Locations (1):
- Dixie Regional Medical Center, Intermountain Healthcare, St. George, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ebell MH, Sokol R, Lee A, Simons C, Early J. How good is the evidence to support primary care practice? Evid Based Med. 2017 Jun;22(3):88-92. doi: 10.1136/ebmed-2017-110704. Epub 2017 May 29. PMID 28554944
- [Background] Berwick DM, Hackbarth AD. Eliminating waste in US health care. JAMA. 2012 Apr 11;307(14):1513-6. doi: 10.1001/jama.2012.362. Epub 2012 Mar 14. PMID 22419800
- [Background] Committee on the Learning Health Care System in America; Institute of Medicine; Smith M, Saunders R, Stuckhardt L, McGinnis JM, editors. Best Care at Lower Cost: The Path to Continuously Learning Health Care in America. Washington (DC): National Academies Press (US); 2013 May 10. Available from http://www.ncbi.nlm.nih.gov/books/NBK207225/ PMID 24901184
- [Background] Special Care Nursery Admissions. (2011). National Perinatal Information Center Quality Analytic Services. Retrieved from https://www.marchofdimes.org/peristats/pdfdocs/nicu_summary_final.pdf
- [Background] Critical Care Statistics. Retrieved from http://www.sccm.org/Communications/Pages/CriticalCareStats.aspx
- [Background] Harrison W, Goodman D. Epidemiologic Trends in Neonatal Intensive Care, 2007-2012. JAMA Pediatr. 2015 Sep;169(9):855-62. doi: 10.1001/jamapediatrics.2015.1305. PMID 26214387
- [Background] National Center for Health Statistics. (2018, January 31). Retrieved from https://www.cdc.gov/nchs/nvss/births.htm
- [Background] Kornhauser M, Schneiderman R. How plans can improve outcomes and cut costs for preterm infant care. Manag Care. 2010 Jan;19(1):28-30. No abstract available. PMID 20131638